CLINICAL TRIAL: NCT02983266
Title: A Study of Safety and Autonomic Responses to Non-Invasive Vagal Stimulation in Persons With Spinal Cord Injury and Non-Disabled Controls Both With and Without Inflammatory Stress
Brief Title: Vagal Nerve Stimulation to Reduce Inflammation and Hyperadrenergia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20150478
Record Dates: First submitted 2016-11-18; First posted 2016-12-06 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Spinal Cord Injury
Keywords: Hyperadrenergia; Inflammatory stress
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (9):
- Group 1: Low Hertz (Experimental): Participants will receive 10 hertz stimulation to the left auricular branch of the vagus nerve, delivered in one 15 minute session.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 1: High Hertz (Experimental): Participants will receive 30 hertz stimulation to the left auricular branch of the vagus nerve, delivered in one 15 minute session.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 1: Control (Sham Comparator): Participants will receive 30 hertz stimulation to a non-vagally innervated region of the left ear, delivered in one 15 minute session.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 2: Pre-stressor (Experimental): Participants will receive 10 or 30 hertz stimulation to the left auricular branch of the vagus nerve, delivered in one 15 minute session prior to receiving experimental sympathetic induction.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 2: Post-stressor (Experimental): Participants will receive 10 or 30 hertz stimulation to the left auricular branch of the vagus nerve, delivered in one 15 minute session after experimental sympathetic induction.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 2: Control (Placebo Comparator): Participants will receive 10 or 30 hertz stimulation to a non-vagally innervated region of the left ear, delivered in one 15 minute session prior to receiving experimental sympathetic induction.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 3: 30 Hz (Experimental): Participants will receive 10 or 30 hertz stimulation to the left auricular branch of the vagus nerve, delivered in one 15 minute session.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 4: 30 Hz (Experimental): Participants will receive 10 or 30 hertz stimulation to the left auricular branch of the vagus nerve, delivered in one 15 minute session. Participants will also receive stimulation on a subsequent session prior to urodynamic testing.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo
- Group 1: Response (Experimental): Participants will receive 10-30 hertz stimulation to the left auricular branch of the vagus nerve, delivered over the course of 1 hour.
  Device: InTENsity MicroCombo
  Interventions: Device: InTENsity MicroCombo

INTERVENTIONS:
Device: InTENsity MicroCombo — An electrotherapy device.

SUMMARY:
The purpose of this research device study is to learn more about the autonomic nervous system. This system uses nerves to send information from the brain to the rest of the body by electrical signaling and has two divisions, the sympathetic and the parasympathetic branches. It has been thought that electrical stimulation devices could be used to restore balance to the nervous system. Because most of the imbalance seems to happen due to too much sympathetic activity, the investigator plans to focus on the parasympathetic branch. Specifically, the investigator hopes to restore balance by targeting the vagus nerve, which is the main communicator of the parasympathetic branch. The study will examine whether the investigator can decrease sympathetic activity and chronic inflammation by increasing parasympathetic activity. This is a device study that will examine the use of non-invasive vagal nerve stimulation to attenuate inflammatory stress and sympathetic hyperactivity in persons with Spinal Cord Injury and Non-Disabled Controls.

ELIGIBILITY:
Group 1 & 2:

Inclusion Criteria:

1. Age 18-65
2. Willingness to participate in the study

Exclusion Criteria:

1. Use of an active electrical implant, such as a cardiac pacemaker or cochlear implant
2. Use of a hearing aid in the left ear
3. Use of an implanted insulin or morphine (pain) pump
4. Self-reported history of syncope from known or unknown origins
5. Self-reported history of cardiovascular disease or dysfunction (e.g., cardiovascular disease, arrhythmia, congestive heart failure, or stroke)

Group 3:

Inclusion Criteria:

1. Age 18-65
2. Overweight, with a BMI ≥ 27
3. Presence of chronic inflammation, with C-reactive protein values > 3 mg/l
4. Willingness to participate in the study

Exclusion Criteria:

1. Use of an active electrical implant, such as a cardiac pacemaker or cochlear implant
2. Use of a hearing aid in the left ear
3. Use of an implanted insulin or morphine (pain) pump
4. Self-reported history of syncope from known or unknown origins
5. Self-reported history of cardiovascular disease or dysfunction (e.g., cardiovascular disease, arrhythmia, congestive heart failure, or stroke)
6. Use of statin drugs

Group 4:

Inclusion Criteria:

1. Age 18-65
2. ≥ 1-year post-injury
3. Bladder management by clean intermittent catheterization
4. Spinal cord injury resulting in Paraplegia level T1 to T6 and motor-complete (AIS A or B) impairment. Injury level and impairment will be confirmed by an ASIA exam conducted less than 2 years before study entry. If longer than 2 years, we will have a certified rater repeat the exam.
5. Participant report of symptoms related to autonomic dysreflexia during episodes of full bladder or voiding, including elevated BP, mild headache, paresthesia, chills, nasal congestion, flushing of the skin, or diaphoresis.
6. Willingness to participate in the study.

Exclusion Criteria:

1. Currently hospitalized
2. American Spinal Injury Association (AIS) C-E
3. Currently using an insulin, morphine (pain), or intrathecal pump
4. Use of an active electrical implant, such as a cardiac pacemaker or cochlear implant
5. Use of a hearing aid in the left ear
6. Self-reported history of syncope from known or unknown origins
7. Self-reported history of cardiovascular disease or dysfunction (e.g., cardiovascular disease, arrhythmia, congestive heart failure, or stroke)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in parasympathetic activity after vagal nerve stimulation by Heart Rate Variability | Baseline to 90 minutes post-vagal nerve stimulation
  Measured by the normal-to-normal QRS complexes of the PQRST waveform of the electrocardiogram (ECG)

SECONDARY OUTCOMES:
Group 1 & 4: Change in acute heart rate response to vagal nerve stimulation | Baseline to 90 minutes post-vagal nerve stimulation
  Measured by numerical heart rate in beats per minute
Group 1 & 4: Change in acute blood pressure response to vagal nerve stimulation | Baseline to 90 minutes post-vagal nerve stimulation
  Measured by diastolic and systolic blood pressure (mm/Hg)
Group 1: Change in parasympathetic activity after vagal nerve stimulation by Vagus Somatosensory Evoked Potentials | Baseline to 90 minutes post-vagal nerve stimulation
  Measured by far field potentials from the brain stem
Group 2 & 4: Change in acute physiological stress response by a change in peripheral cortisol | Baseline to 90 minutes post-experimental stimulus
  Measured by cortisol levels in plasma
Group 2 & 4: Change in acute physiological stress response by a change in peripheral catecholamines | Baseline to 90 minutes post-experimental stimulus
  Measured by catecholamine levels in plasma
Group 2 & 4: Change in acute physiological stress response by a change in heart rate | Baseline to 90 minutes post-experimental stimulus
  Measured by numerical heart rate in beats per minute
Group 2 & 4: Change in acute physiological stress response by a change in blood pressure | Baseline to 90 minutes post-experimental stimulus
  Measured by diastolic and systolic blood pressure (mm/Hg)
Group 3 & 4: Change in inflammatory biomarkers after vagal nerve stimulation | Baseline to 90 minutes post-vagal nerve stimulation
  Measured by cytokine levels in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, Ph.D., Principal Investigator — University of Miami
Locations (1):
- The Miami Project to Cure Paralysis/ University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No